CLINICAL TRIAL: NCT04568239
Title: Impact of M184V on the Virological Efficacy to Lamivudine/Dolutegravir
Brief Title: Impact of M184V on the Virological Efficacy to 3TC/DTG (LAMRES)
Acronym: LAMRES
Status: Completed | Type: Observational
Sponsor: Association de Recherche en Virologie et Dermatologie (Other)
Responsible Party: Sponsor
Other Study IDs: ARVD-LAMRES
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- M184V + group and M184 - group

SUMMARY:
In view of the prolongation of patients living with HIV's life expectancy, the question of optimization of ART, which is still a life-long treatment, becomes central. While most patients achieve virological success, their treatments often need to be optimized in order to limit adverse events, drugs interactions and to improve adherence. The switch to dual regimen strategies represent one of the approaches for treatment optimization. Indeed, dual therapy regimens have shown non-inferior efficacy vs triple therapy as simplification therapy and more recently also as first line therapy. From the real-life data it emerges that today in simplification strategies, the dual regimen therapies are prescribed even in patients with a history of virological failure. Circulating HIV-1 resistant variants can be archived in viral reservoirs, where they can persist for years and can reemerge in case of therapeutic selective pressure. In particular, previous selection of M184V may have an impact on virological response to 3TC/DTG. There are few data on a direct comparison of 3TC/DTG efficacy in patients harboring or not harboring the M184V. So, there is a need to assess the efficacy of 3TC/DTG in patients with past M184V mutation in a large set of patients followed in clinical setting.

Thus, the investigators propose a retrospective study of patients with HIV-RNA ≤50 copies/mL who were switched to 3TC/DTG in order to compare the virological efficacy of 3TC/DTG in patients with and without a history of M184V detection in a previous resistance genotype. This study aimed to analyze 800 patients switched to DTG/3TC in clinical real setting in large European (France, Italy, Spain) database.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Age ≥ 18 years
* Switched to 3TC/DTG while having HIV-RNA ≤50 copies/mL on any ART regimen
* Followed for at least 1 year after 3TC/DTG switch
* With at least 1 previous genotype
* With at least 1 virological follow-up after switching to 3TC/DTG

Exclusion Criteria:

* No genotypic resistance test available before switching to DTG/3TC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1-infected patients with (i) age ≥18 years, (ii) HIV-RNA ≤50 copies/mL on any ART regimen, (iii) subsequently switching to DTG/3TC, (iv) with at least 1 previous plasma HIV-1 RNA or HIV-DNA genotype, (v) with at least 1 virological and clinical follow-up after switching to DTG/3TC.
  The occurrence of M184V will be assessed using historical genotypic resistance tests; that is, any detection of this mutation in any previous resistance test will be scored as positive.
Sampling Method: Non-Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
probability of virological failure | 12 months
  probability of virological failure that is defined as HIV-RNA >50 copies/mL in 2 consecutive determinations or ≥200 copies/mL in a single determination. This outcome will be evaluated overall and between the M184V- and M184V+ patients' groups.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Genevieve Marcelin, PharmD, PhD, Principal Investigator — Sorbonne University; APHP
Locations (1):
- ARVD, Paris, France